CLINICAL TRIAL: NCT01123902
Title: Effectiveness of a Hand-held Fan for Breathlessness: a Randomised Phase II Trial
Brief Title: Effectiveness of a Hand-held Fan for Breathlessness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Prof Irene Higginson, King's College London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CREC 05/06-69
Record Dates: First submitted 2010-05-11; First posted 2010-05-14 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2006-07

CONDITIONS: Primary Lung Cancer or Secondary Lung Metastases; COPD III/IV
Keywords: Breathlessness; Dyspnea; Hand-held fan; Palliative Care
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hand-held fan (Experimental)
  Interventions: Device: hand-held fan
- wristband (Placebo Comparator)
  Interventions: Device: wristband

INTERVENTIONS:
Device: hand-held fan — Patients are instructed to direct the hand-held fan towards the face around the central part of the face, the sides of the nose and above the upper lip. The hand-held fan has three soft rotor blades and an unfoldable rotor unit.
  Arms: hand-held fan
Device: wristband — Patients are instructed to wear the wristband continually and pull it regularly at short intervals when breathless or during breathlessness attacks.
  Arms: wristband

SUMMARY:
Breathlessness is a common and distressing symptom in advanced disease. A hand-held fan is a simple device which has shown, when directed to the patients face, to be effective in relieving breathlessness.

This phase II trial aims to determine the potential effectiveness of a hand-held fan to relieve breathlessness over time and to evaluate the recruitment into the study and the acceptance of the intervention and the control.

The intervention to be tested is a HHF directed to the area of the face innervated by the second and third trigeminal nerve branches. A wristband was chosen as control under the assumption that distraction could serve as a placebo.

The main outcomes for this study are uptake into the trial (proportion of patients from the longitudinal study participating in the RCT), adherence to the study, and use and acceptance of the intervention and the control. The main outcome for assessing the effect of the hand-held fan is change of severity of breathlessness between baseline and one month and two months, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients were included if they reported breathlessness that had an impact on their daily life and were suffering from one of the following conditions:
* Advanced malignant disease (primary lung cancer or secondary lung metastases/ lung involvement due to cancer)
* COPD stage III (severe) and IV (very severe) according to GOLD criteria.[7]

Exclusion Criteria:

* Unable to provide informed consent
* Too ill to be interviewed and not fluent or illiterate in German

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2006-06; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
change of severity of breathlessness | between baseline and one month

SECONDARY OUTCOMES:
use and acceptance of the intervention and the control | over 6 months
adherence to the study | 6 months
uptake into the trial (proportion of patients from the longitudinal study participating in the RCT) | 18 months
change of severity of breathlessness | baseline and two months

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Bausewein, PhD MD MSc, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

REFERENCES:
- [Derived] Bausewein C, Booth S, Gysels M, Kuhnbach R, Higginson IJ. Effectiveness of a hand-held fan for breathlessness: a randomised phase II trial. BMC Palliat Care. 2010 Oct 19;9:22. doi: 10.1186/1472-684X-9-22. PMID 20958972